CLINICAL TRIAL: NCT02853994
Title: Assessment of Safety and Efficacy of the DEVOIR Sirolimus-Coated Balloon for the Treatment of Native Coronary Artery Lesions in the Real-world Clinical Practice
Brief Title: Safety and Efficacy of the DEVOIR Sirolimus-Coated Coronary Balloon in the Real-world Clinical Practice
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: MINVASYS (Industry)
Responsible Party: Sponsor
Other Study IDs: P1601
Record Dates: First submitted 2016-07-18; First posted 2016-08-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-07

CONDITIONS: CAD
Keywords: DCB; DEB; Sirolimus; PCI; ISR; SVD; Restenosis; Bifurcation; CAD; Coronary artery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study is a prospective, non-randomized, multicenter, post-marketing surveillance study evaluating the CE-marked DEVOIR Sirolimus-Coated Coronary Balloon in 4 subgroups regarding device approved indications:

* In-stent restenosis lesions: either bare metal or drug eluting stent restenosis
* Bifurcation lesions (with drug-eluting stent in main branch and drug-coated balloon in side branch): treatment of lesion of all Medina types except (0,0,1) in native coronary arteries
* Small vessels: treatment of lesions ≤2.75 mm
* BMS implantation followed by DCB inflation

ELIGIBILITY:
Patient's inclusion and exclusion criteria are per device instructions for use's indications and contraindications.

Inclusion criteria:

1. Patient is at least 18 years old
2. Lesion lengths ranging from 8 to 38 mm and diameters ranging from 1.50 mm to 4.00 mm.

Exclusion criteria:

1. Patients with a hypersensitivity to Sirolimus drug or its structural activity related compounds.
2. Patients with a known hypersensitivity to excipients with phospholipid or related origins.
3. Patients whose diseased segment cannot be pre-dilated or prepared before drug coated balloon treatment.
4. Severely calcified lesions requiring treatment of other type for e.g. Rotational Atherectomy (Rotablator)
5. Patients judged to have lesion that prevents complete inflation of angioplasty balloon or proper placement of delivery catheter
6. Patients who cannot receive recommended antiplatelet or anticoagulation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery diseases (in-stent restenosis, small vessel diseases, bifurcation lesions, de novo lesions)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Rate of Major Adverse Cardiac Events (MACE) | 12 months

SECONDARY OUTCOMES:
Rate of Target Lesion Revascularization (TLR) | 12 months
Rate of Target Vessel Failure (TVF) | 12 months
Rate of Target Vessel Revascularization (TVR) | 12 months
Angiographic success | Day 1